CLINICAL TRIAL: NCT02424292
Title: Evaluating the Outcome of a Personalised Oncological Rehabilitation Program in Overweight and Obese Breast Cancer Patients on Adjuvant Anti-hormonal Treatment "I-Move"
Brief Title: Evaluation of a Physical Activity Program in Overweight Breast Cancer Patients
Acronym: I-Move
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Pink Ribbon Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: I-Move; NL44459.042.13 (Other: ABR form)
Record Dates: First submitted 2015-04-13; First posted 2015-04-23 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Physcial activity/exercise; anti-hormonal treatment
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Physical activity: Physical activity in a personalised program
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — Physical activity in a personalised program.

SUMMARY:
Patients diagnosed with breast cancer generally have a fairly well prognosis with estimated average survival rates of 73% and five year survival rates of 89% in developed countries. However, women who are obese at the time of breast cancer diagnosis seem to be at risk for a worse breast cancer related and overall survival, as compared to their normal weight counterparts. In addition, weight gain after diagnosis might be negatively associated with prognosis.

Weight gain is a common phenomenon among breast cancer patients receiving adjuvant chemotherapy as well as receiving adjuvant anti-hormonal therapy. While sufficient physical activity and limitation of the amount of weight gain is important for all breast cancer patients, it surely is for overweight and obese patients. The recently published national guideline oncological rehabilitation provides exercise goals, for physical training based on the Dutch PA guideline "Nederlandse Norm Gezond Bewegen (NNGB)". It recommends to engage in moderate-intensity exercise (e.g. brisk walking) for at least 30 minutes a day, on at least 5 days a week. For people who are overweight (Body Mass Index ≥ 25 kg/m2) it is recommended to exercise at least 60 minutes at a moderate-intensity level, equal or more than 3 Metabolic Equivalent Task Hours (> 3 MET/h), on at least 5 days a week. However, only 61% of the general population, meets these guidelines (8) and among cancer patients this percentage is even less. This study aims to increase the percentage of overweight breast cancer patients treated with adjuvant anti-hormonal therapy that reaches the goal of the NNGB by the oncological rehabilitation program with 20%.

DETAILED DESCRIPTION:
Rationale:

Patients diagnosed with breast cancer generally have a fairly well prognosis with estimated average survival rates of 73% and five year survival rates of 89% in developed countries (1). However, women who are obese at the time of breast cancer diagnosis seem to be at risk for a worse breast cancer related and overall survival, as compared to their normal weight counterparts. In addition, weight gain after diagnosis might be negatively associated with prognosis. Possible mechanisms explaining this association include host-related, tumour-related and treatment-related factors (2).

Regular physical activity (PA) after a diagnosis of breast cancer can have various beneficial effects with respect to overall survival (3) as well as health-related quality of life (4). The Dutch PA guideline "Nederlandse Norm Gezond Bewegen (NNGB)" recommends to engage in moderate-intensity exercise (e.g. brisk walking) for at least 30 minutes a day, on at least 5 days a week (5). For people who are overweight (Body Mass Index ≥ 25 kg/m2) it is recommended to exercise at least 60 minutes at a moderate-intensity level, equal or more than 3 Metabolic Equivalent Task Hours (> 3 MET/h), on at least 5 days a week (6,7). However, only 61% of the general population, meets these guidelines (8) and among cancer patients this percentage is even less (9).

The recently published national guideline oncological rehabilitation provides exercise goals, for physical training based on the NNGB (5) as well as advice regarding nutrition and education on maintaining a healthy lifestyle. The guideline emphasises the importance of a tailored program, taking into account personal preferences and attitudes concerning physical exercise. Level of PA self-efficacy (beliefs in one's capabilities to successfully execute the required PA) is mentioned as an important predictor of compliance.

Weight gain is a common phenomenon among breast cancer patients receiving adjuvant chemotherapy (10) as well as receiving adjuvant anti-hormonal therapy (11). While sufficient physical activity and limitation of the amount of weight gain is important for all breast cancer patients, it surely is for overweight and obese patients. In the provinces of Groningen and Drenthe, the percentage of overweight women is significantly higher compared to the national average. In addition, in this area the average socio-economic status (SES), often associated with unhealthy lifestyle, overweight and not seeing the personal relevance of health recommendations, is lower than in the rest of the Netherlands. This leaves this group extra vulnerable for all kinds of health problems like diabetes mellitus, hypertension, increased risk of cardiovascular disease and decreased cancer related survival. However, it is also known to be a population that is very difficult to motivate to engage in more physical activity. Therefore, it is uncertain if the guideline oncological rehabilitation is sufficient enough to reach the NNGB goals. Oncological rehabilitation can render health gain in this patient population, as it can potentially limit weight gain, improve parameters of metabolic syndrome and improve health-related quality of life.

Objective: To increase the percentage of overweight breast cancer patients treated with adjuvant anti-hormonal therapy that reaches the goal of the NNGB by the oncological rehabilitation program with 20%.

Secondary objectives: To evaluate whether the possible increase in percentage of patients meeting the NNGB is sustained up to 26 weeks (=3 months) after completion of the oncological rehabilitation. To evaluate the effect of oncological rehabilitation on body composition including weight, on parameters of metabolic syndrome, on health-related quality of life and on self-efficacy in this patient population.

Study design: The primary aim of this study is to determine whether oncological rehabilitation results in reaching the goals of the NNGB for overweight breast cancer patients. A single-arm, experimental pre-post test design, evaluating preliminary effectiveness of a 12-week personalised oncological rehabilitation program in overweight or obese (BMI ≥ 25 kg/m2) breast cancer patients, on adjuvant anti-hormonal therapy will be used. The oncological rehabilitation program will vary according to patients' baseline characteristics, possible functional limitations and personal preferences. Assessment of meeting the NNGB (by accelerometry), of body composition, parameters of metabolic syndrome, health-related quality of life and self-efficacy, will be performed at baseline, immediately after completion of the 12 week study period and at follow-up 26 weeks after baseline (= 3 months after completion of the intervention). Changes in these parameters between baseline and 12 weeks and baseline and 26 weeks will be analysed. The secondary aims are to establish the effect of physical activity on the prevalence of metabolic syndrome, the quality of life and self-efficacy in this group of patients. These secondary parameters will be assessed as a positive reinforcement for patients to continue with the engaged physical activities.

Study population: 141 overweight or obese (BMI ≥ 25 kg/m2) women 18-75 years old who are treated with adjuvant anti-hormonal therapy for breast cancer.

Intervention: Patients will be offered a personalised program following the guidelines of oncological rehabilitation, which over a period of 12 weeks will facilitate them to stepwise increase the level of PA up to meeting the PA guideline for overweight/obese people. To explore physical activity patients will be asked to wear an accelerometer during 1 week before the start of the oncology rehabilitation program (baseline). For patients already meeting the guideline at baseline, the program will stimulate them to keep doing so and other aspects of achieving a healthy lifestyle will be discussed together with the physiotherapist.

Hereto all patients will have an intake with the physiotherapist of the oncology rehabilitation program assessing personal preferences with regard to physical activities, hindering factors as well as functional limitations in the individual patient. Possible solutions for hindering factors will be sought for. Based on patient's individual characteristics and preferences, the physiotherapist will create a tailored PA program for this individual patient to stimulate them in meeting the PA guidelines at the end of the study period. To facilitate meeting the guidelines, patients can follow a supervised PA program (individual or group-wise) 2-3 times a week, or a combination of an unsupervised home-based program (individual or group-wise) with a supervised program. Activities engaged will be gradually increased in duration per session and/or intensity. In addition, incorporating physical activity in the daily routine (household activities, going to the shop by bike instead of by car) will be stimulated. All patients will have follow-up conversations by skype/facetime or telephone after 1, 3 and 7 weeks.

Evaluation of the set goals, of possible hindering factors and how to overcome them, encouragement and - if needed and in consultation with the physiotherapist - setting new realistic goals for the next period will be standard part of these follow-up conversations.

Main study parameters/endpoints:

Primary endpoint:

The percentage of patients meeting the Dutch PA guideline for overweight/obese people (≥ times one hour per week) after completion of the 12 week intervention. Meeting the guideline will be measured with accelerometry (12).

Secondary endpoints:

* Sustainability of the possible increase in percentage of patients meeting the Dutch PA guideline for overweight or obese people up to 3 months after completion of the intervention.
* Changes in body composition (weight, BMI, fat percentage as measured with the skinfold measurements), parameters of metabolic syndrome (waist circumference, blood pressure, fasting blood glucose, high density lipoprotein, triglycerides), health-related quality of life (using EORTC QLQ-C30, the EORTC BR23 and single question on satisfaction with life) and general and PA self-efficacy (using the ALCOS and PA self-efficacy questionnaire respectively), between baseline,12 weeks after baseline and 26 weeks thereafter.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Despite participation in this study being reserved for those without any contra-indication for physical exercise and despite the conclusion of the American College of Sports Medicine Roundtable on Exercise Guidelines for Cancer Survivors that exercise is safe during and after cancer treatment (13), in doing physical exercise there is always a risk of (sports) strain/injury. However, regarding the nature of the targeted intensity of exercise (moderate), this risk will be low and the investigators expect the benefits (both physically and psychologically) to far outweigh possible risks.

At baseline and 12 and 26 weeks thereafter, the following assessments will be performed: measurement of physical activity with an accelerometer, measurement of body composition (weight, BMI, fat percentage as measured with the skinfold measurements), parameters of metabolic syndrome (this includes measuring waist circumference and blood pressure, drawing blood to measure fasting blood glucose, high density lipoprotein and triglycerides). In addition, filling out questionnaires on general physical activity (ALCOS) and PA self-efficacy (PA self-efficacy questionnaire), health-related quality of life including satisfaction (EORTC QLQ-C30, the EORTC BR23 and single question on satisfaction with life) will be part of the study. Information on these questionnaires can be found in Appendix 5.

At baseline, a questionnaire regarding baseline characteristics (marital status, education level, employment status, monthly household income, being advised to exercise by the treating oncologist, being on a diet with the purpose of losing weight, known with diabetes, hypertension, hypercholesterolemia, current medication and stage of behavioural change) will be filled out. Medical record will be viewed by the researcher for additional patient characteristics like tumour stage at diagnosis (see 5.1.3).

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients
* Diagnosis of stage I-III breast cancer, currently on adjuvant anti-hormonal treatment
* BMI ≥ 25 kg/m2
* Age 18-75 years old
* Provided informed consent

Exclusion Criteria:

* Evidence of recurrent/metastatic breast cancer or other primary malignancy
* Uncontrolled heart disease
* Other contraindications to exercise training (e.g., orthopaedic problems)
* Dementia

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female breast cancer patients treated with hormonal therapy in adjuvant setting and a BMI≥ 25 kg/m2
Sampling Method: Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2015-04; Primary Completion 2019-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Measure by accelerometry whether patients meet Dutch PA guidelines for overweight/obese people. | 12 weeks
  measured in minutes per week >3 METs was attained

SECONDARY OUTCOMES:
Measure whether possible change in physical activity is sustained up to 3 months. | 26 weeks
  measured in minutes per week >3 MET was attained

CONTACTS AND LOCATIONS:
Overall Officials: A. KL Reyners, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (4):
- Netherlands (4):
  - Wilhelmina Ziekenhuis, Assen
  - Martini Ziekenhuis, Groningen
  - UMCG, Groningen
  - OZG, Winschoten

REFERENCES:
- [Derived] Ormel HL, Schroder CP, van der Schoot GGF, Westerink NL, van der Velden AWG, Poppema B, Vrieling AH, Gietema JA, Walenkamp AME, Reyners AKL. Effects of supervised exercise during adjuvant endocrine therapy in overweight or obese patients with breast cancer: The I-MOVE study. Breast. 2021 Aug;58:138-146. doi: 10.1016/j.breast.2021.05.004. Epub 2021 May 15. PMID 34023558